CLINICAL TRIAL: NCT04851145
Title: Diagnostic Value of Mass Spectrometry-based Proteomics in Microvascular Inflammation in Kidney Transplantation, the TranSpec Study.
Brief Title: Mass Spectrometry-based Proteomics in Microvascular Inflammation Diagnosis in Kidney Transplantation.
Acronym: TranSpec
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/47
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplantation; Graft Rejection; Humoral Immunity; Proteomics
Keywords: Antibody-mediated rejection; microvascular inflammation; proteomics; kidney transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Diagnostic Test: Mass spectrometry-based proteomics of FFPE biopsies and urine samples

INTERVENTIONS:
Diagnostic Test: Mass spectrometry-based proteomics of FFPE biopsies and urine samples — The biopsy and urine samples will be processed by the OncoProt platform (University of Bordeaux) for proteomic analysis by tandem mass spectrometry (label-free quantification) as follows:
  * Biopsies: laser microdissection of the renal cortex, fixation reversion, protein extraction and electrophoretic migration, tryptic digestion.
  * Urines: samples concentration by centrifugation/filtration and tryptic digestion according to a protocol adapted from the FASP method (Filter-Aided Sample Preparation)

SUMMARY:
Microvascular inflammation, the hallmark histological criteria of antibody-mediated rejection in kidney transplantation, remains an issue in routine practice, due to a lack of reproducibility in its recognition by pathologists and an incomplete comprehension of its pathophysiology, leading to a poor treatment efficacy. The main objective of this study is to assess the performances of tissue proteic signatures designed for the diagnosis of microvascular inflammation in kidney transplantation, from formalin-fixed and paraffin-embedded (FFPE) allograft biopsies analyzed by mass spectrometry-based proteomics.

DETAILED DESCRIPTION:
Antibody-mediated rejection (ABMR) is due to pathogenic antibodies produced by the donor (donor-specific antibodies, DSA) that are directed against Human Leukocyte Antigens (HLA) or other antigens (non HLA) of the graft. ABMR is currently the leading cause of long-term kidney allograft failure. Histological lesions of microvascular inflammation (MVI) are the hallmark criteria of ABMR according to the 2019 Banff classification. Lack of reproducibility in the scoring of MVI by pathologists is still an issue of the diagnosis of ABMR in routine practice, while the understood pathophysiological mechanisms of MVI (anti-HLA DSA, DSA against non HLA antigens and/or NK cell-mediated) are poorly assessed in practice, possibly explaining the wide variability of treatment efficacy. In a prior study, the investigators confirmed the value of mass spectrometry for the analysis of the glomerular proteome during ABMR, compared to the one of stable grafts, from FFPE biopsies. The investigators identified 82 proteins, particularly involved in leukocyte activation and the interferons pathways, in accordance with transcriptomic approaches. Five proteins were validated by immunohistochemistry.

The investigators now propose to analyze kidney allograft FFPE biopsies of 92 patients by mass spectrometry, including 32 with MVI (with and without anti-HLA DSA) and 60 with relevant differential diagnoses. The main objective is to assess the diagnostic performances of tissue proteic signatures designed by machine-learning methods for the diagnosis of microvascular inflammation, the reference standard being the 2019 Banff classification. One of the secondary objectives includes the comparison of the protein profile of MVI with and without anti-HLA DSA, but also the proteomic analysis of 60 urine samples from the same population, in order to assess the performances of mass spectrometry in the non-invasive diagnosis of MVI in kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* Diagnosis based on the 2019 Banff classification (polyomavirus nephropathy, T cell-mediated rejection, borderline changes)
* Renal allograft biopsy allowing inclusion with at least 7 permeable glomeruli
* The microvascular inflammation group with anti-HLA DSA is defined as follows:

  * At least moderate microvascular inflammation: g + ptc > 2
  * At least one anti-HLA DSA in the serum at the time of biopsy, with a Mean Fluorescence Intensity (MFI) > 3000 for the immunodominant DSA or the sum of the DSA
* The microvascular inflammation group without anti-HLA DSA is defined as follows:

  * At least moderate microvascular inflammation: g + ptc > 2
  * No historical anti-HLA DSA or at the time of biopsy, MFI < 500
* The stable graft recipients group is defined as follows:

  * Glomerual Filtration Rate > 40ml/min, without clinical proteinuria
  * No detectable DSA
  * Protocol biopsy at 1 year posttransplantation without specific lesion or nonspecific severe lesion
* The chronic nonspecific graft changes group is defined as follows:

  * Moderate to severe interstitial fibrosis and tubular atrophy, in the absence of specific lesions: active rejection (antibody-mediated or T cell-mediated), borderline lesions, recurrent or de novo nephropathy, polyomavirus associated nephropathy.
  * No C4d deposits on peritubular capillaries
  * No detectable anti-HLA DSA at the time of biopsy.
* The ischemic acute tubular injuries group is defined as :

  * Histological lesions of tubular injuries in the absence of significant microvascular inflammation or C4d deposits
  * No detectable anti-HLA DSA at the time of biopsy

Exclusion Criteria:

* Minor patients
* Mixed rejection (antibody-mediated and T cell-mediated)
* Recurrent or de novo nephropathy
* Specific treatment of rejection (T cell-mediated or antibody-mediated) in the last 6 months, excluding induction and
* Baseline immunosuppressive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Assessing diagnostic performance of tissue protein signature | 18 months after inclusion
  The primary outcome is the sensitivity and specificity of tissue protein signature in the diagnosis of microvascular inflammation (MVI) in kidney transplantation, the diagnostic reference standard being based on the 2019 Banff classification (histological and biological criteria). This primary outcome is based on FFPE kidney allograft biopsies.

SECONDARY OUTCOMES:
Assessing the diagnostic performance of urine protein signatures | 18 months after inclusion
  Sensitivity and specificity of the urinary protein signature in the diagnosis of MVI in kidney transplantation, compared to the reference standard (2019 Banff classification)
Assessing the performance of tissue proteomic signature | 18 months after inclusion
  Sensitivity and specificity of tissue proteomic analysis in the prediction of the MVI subtype (anti-HLA DSA or not)
Assessing the performance of urine proteomic signature | 18 months after inclusion
  Sensitivity and specificity of urine proteomic analysis in the prediction of the MVI subtype (anti-HLA DSA or not)
Compare protein profiles observed within different phenotypes of MVI in kidney transplantation | 18 months after inclusion
  To describe and compare protein profiles observed within different phenotypes of MVI in kidney transplantation, at tissue and urine protein level according to Banff 2019 (with and without anti-HLA DSA).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Necker, Paris

IPD SHARING:
Plan to Share IPD: No